CLINICAL TRIAL: NCT02757170
Title: Assessment of Coagulation Abnormalities in Acute on Chronic Liver Failure Patients Using Thromboelastography
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Subrat Kumar Acharya, Professor, Department of Gastroenterology, All India Institute of Medical Sciences
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: IESC/T-203/05.05.15
Record Dates: First submitted 2016-04-25; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Acute on Chronic Liver Failure; Cirrhosis
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Fibrosis | interventions — Thrombelastography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- I (Experimental): Thromboelastography Acute on chronic liver failure: Patients' whole blood will be taken and subjected to undergo coagulation with thromboelastometry and various graphic tracings will be recorded which will highlight the process of coagulation in these patients
  Interventions: Device: Thromboelastography
- Group II (Active Comparator): Thromboelastography Healthy Controls: Healthy persons' whole blood will be taken and subjected to undergo coagulation with thromboelastometry and various graphic tracings will be recorded which will highlight the process of coagulation.
  Interventions: Device: Thromboelastography
- Group III (Experimental): Thromboelastography Chronic Liver Failure: Patients' whole blood will be taken and subjected to undergo coagulation with thromboelastometry and various graphic tracings will be recorded which will highlight the process of coagulation in these patients
  Interventions: Device: Thromboelastography
- Group IV (Experimental): Thromboelastography Acute Liver Failure: Patients' whole blood will be taken and subjected to undergo coagulation with thromboelastometry and various graphic tracings will be recorded which will highlight the process of coagulation in these patients
  Interventions: Device: Thromboelastography

INTERVENTIONS:
Device: Thromboelastography — Patients whole blood will be subjected to undergo coagulation process under monitoring with thromboelastography and various tracings will be recorded and will be interpreted as results.

SUMMARY:
Patients of acute & chronic liver failure have long been assumed to have coagulopathy & are given blood products prophylactically as well as during various interventions. But these patients rarely have spontaneous bleed except variceal bleed. Conventional coagulation parameters are insufficient to assess coagulation status of these patients because they reflect only a certain element of coagulation cascade while thromboelastography (TEG) gives a comprehensive report of hemostatic profile including platelet function. Studies using TEG have suggested that defects in prohemostatic drivers are counterbalanced by changes in antihemostatic drivers creating a rebalance in these patients. Acute on chronic failure is a entity with acute decompensation on underlying chronic liver failure. Since there is paucity of data regarding coagulation abnormalities in these patient, study is needed to assess predictability power of TEG in these patients with respect to coagulation abnormalities in patient with ALF and CLD ( cirrhosis) and healthy controls.

DETAILED DESCRIPTION:
Since early times coagulopathy is considered to be an integral part of liver failure. Whether it is acute liver failure (ALF) or acute on chronic liver failure (ACLF), patients usually have deranged coagulation parameters (platelet count, prothrombin time (PT), activated partial thromboplastin time (aPTT) and international normalized ratio (INR). Based on these deranged parameters, initially it was assumed that patients of liver failure have increased risk of bleeding & usually were given blood products prophylactically during surgical interventions. But these patients of liver failure (acute or chronic) seldom develop spontaneous bleeding, apart from variceal bleeding in chronic liver failure which generally occurs because of portal hypertension. Moreover during invasive procedures also they do not have significant bleeding.

Concept of rebalanced hemostasis has been proposed to explain discrepancy between results of these coagulation parameters & clinical scenario of patients. Normal hemostasis consists of 3 steps: platelet endothelial interaction, coagulation & fibrinolysis. First step is considered to be defective in liver failure because of thrombocytopenia & qualitative platelet dysfunction. However because of decreased plasma concentration of ADAMTS 13, plasma levels of vwF are increased thus increasing stickiness of platelets & rebalancing the primary hemostasis.

Because of deranged INR, it is thought that coagulation cascade is deranged but Tripodi et al have shown that cirrhotics also can generate same amount of thrombin as healthy subjects. All procoagulants (factor II, V, VII, IX, X, XI) & anticoagulant factors (protein C, protein S & antithrombin) except factor VIII are synthesized in liver. Decreased procoagulant activity has been found to be counterbalanced by decreased anticoagulant proteins, thus rebalancing the whole coagulation process.

Finally, there is increased fibrinolytic activity and clot instability because of increased tissue plasminogen activator (tPA) with low levels of alpha 2 antiplasmin, factor XIII and reduced thrombin activated fibrinolysis inhibitor (TAFI). However, this is balanced by increased levels of acute phase reactant plasminogen activator inhibitor (PAI-1).

Conventional parameters like INR although can predict mortality in these cases but don't predict risk of bleeding in these patients because they monitor only a part of coagulation cascade. These parameters assess clot formation in plasma environment while in Thromboelastography (TEG) whole blood i.e. both plasma & cellular components including platelets are assessed & a collective report of hemostatic profile of patient is available. Graph obtained using TEG gives 5 values including r time, k time, α angle, maximum amplitude & lysis at 30 min assessing different aspects. It has been widely used prior to cardiac surgery and liver transplant surgery to assess for coagulation defects.

In patients with stable cirrhosis, the TEG parameters are reported to lie within normal limits. TEG measurements done serially have been shown to be better than routine coagulation tests in measuring hypocoagulability in cirrhotics with early rebleeding. In decompensated cirrhotic patients, bacterial infections are common and impair hemostasis. The TEG parameters are impaired on the day of infection and recover to normal values in 5 days in cases showing response to treatment.

The results of TEG in ALF have been contrasting in the two studies which included predominantly paracetamol induced ALF. Stravitz et al in a study of 51 ALF patients reported normal TEG in 63%, 1 abnormality in 16%, 2 abnormalities in 10%, 3 abnormalities in 8% of patients and 4 abnormalities in 4% whereas 8% patients had TEG parameters in a hypercoagulable range though the mean of parameters were within normal limits in all patients. In another study of 20 ALF patients, TEG findings were consistent with a hypocoagulable state in 20%, normal in 45%, and hypercoagulable in 35% of the patients.

Acute on chronic liver failure is a recently defined entity with prolonged INR being a component of definition. The exact nature of coagulopathy in this disease has not yet been studied. In this prospective study, we propose to study the role of TEG in assessing the coagulation state in patients with ACLF and comparing the TEG parameters with respect to patients with ALF, CLD and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive ALF, ACLF & cirrhotic patients and healthy controls
2. Written informed consent (patient or his nearest relative)

Exclusion Criteria:

1. Patients on anti-platelet or anticoagulant therapy
2. Pregnancy and immediate post-partum period
3. History of underlying hypercoagulable/ hypocoagulable states eg. PNH, Polycythemia, Hemophilia
4. Patients with renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Changes in r, k and MA- TEG parameters in ACLF | 1 day

SECONDARY OUTCOMES:
Comparison of r, k and MA- TEG parameters with conventional tests of coagulation (i.e PT, aPTT) | 1 day
Development of renal failure, progression of hepatic encephalopathy, variceal bleeding and sepsis in patients with r, k and MA- TEG parameters | 28 days
Death in patients with abnormal r, k and MA- TEG parameters | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Subrat k Acharya, DM, Principal Investigator — AIIMS, New Delhi
Locations (1):
- Dr. S K Acharya, New Delhi, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided